CLINICAL TRIAL: NCT00836693
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Assess the Efficacy and Safety of Tadalafil (LY450190) Once a Day in Subjects With Erectile Dysfunction Who Are Naïve to PDE5 Inhibitors
Brief Title: Effect of Tadalafil Once a Day in Men With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12229; H6D-MC-LVHX (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental)
  Interventions: Drug: tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tadalafil — 5 milligrams (mg) administered orally once a day for 12 weeks
  Other Names: Cialis; LY450190
  Arms: Tadalafil
Drug: placebo — tablet administered orally once a day for 12 weeks.
  Arms: Placebo

SUMMARY:
The primary aim of this study is to assess the efficacy and safety of tadalafil 5 mg administered once a day in patients with erectile dysfunction (ED) who are naïve to PDE5 (phosphodiesterase type 5) inhibitors. Patients may be dose reduced to 2.5mg based on tolerability.

ELIGIBILITY:
Inclusion Criteria:

* You are male and aged at least 18 years.
* Have a history of erectile dysfunction (ED)(defined as the consistent inability to achieve and/or maintain an erection sufficient to permit satisfactory sexual intercourse) of at least 3 months duration.
* Agree not to use any other treatment for ED, including herbal and over-the-counter (OTC) medications, during the study
* You agree to make at least four sexual intercourse attempts with the female sexual study partner during the 4-week run-in period without medication
* Your entry laboratory test results and medical tests meet study requirements
* You agree to use the study drug only as instructed by your study doctor and staff and to return any unused study drug and containers at the end of the study or as otherwise instructed by the study doctor.
* If currently using cholesterol lowering medications (for example: statins) or medications to lower blood pressure (example: angiotensin-converting enzyme (ACE) inhibitors or calcium channel blocker medications), you need to be on a stable dose and you and your study doctor do not expect any dose change during the study.

Exclusion Criteria:

* You have received previous or current treatment with tadalafil or any other PDE5 inhibitor.
* Currently receives treatment with doxazosin, nitrates, cancer chemotherapy, or anti-androgens (except finasteride e.g. Propecia™ or Proscar®, or dutasteride e.g. Avodart®).
* You have had significant heart disease as determined by your doctor in charge of this study or a member of the doctor's staff.
* Have a history of significant central nervous system injuries (including stroke or spinal cord injury) within the last 6 months.
* Have a history of loss of vision in one eye because of nonarteritic anterior ischemic optic neuropathy (NAION), regardless of whether this episode was in connection or not with previous PDE5 inhibitor exposure.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-459) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Wiessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Koblenz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., L’Aquila
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Legionowo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aravaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Majadahonda

REFERENCES:
- [Derived] Porst H, Gacci M, Buttner H, Henneges C, Boess F. Tadalafil once daily in men with erectile dysfunction: an integrated analysis of data obtained from 1913 patients from six randomized, double-blind, placebo-controlled, clinical studies. Eur Urol. 2014 Feb;65(2):455-64. doi: 10.1016/j.eururo.2013.09.037. Epub 2013 Oct 2. PMID 24119319
- [Derived] Porst H, Brock GB, Kula K, Moncada I, Montorsi F, Basson BR, Kinchen K, Aversa A. Effects of once-daily tadalafil on treatment satisfaction, psychosocial outcomes, spontaneous erections, and measures of endothelial function in men with erectile dysfunction but naive to phosphodiesterase type 5 inhibitors. J Androl. 2012 Nov-Dec;33(6):1305-22. doi: 10.2164/jandrol.111.015289. Epub 2012 Jul 12. PMID 22790642
- [Derived] Montorsi F, Aversa A, Moncada I, Perimenis P, Porst H, Barker C, Shane MA, Sorsaburu S. A randomized, double-blind, placebo-controlled, parallel study to assess the efficacy and safety of once-a-day tadalafil in men with erectile dysfunction who are naive to PDE5 inhibitors. J Sex Med. 2011 Sep;8(9):2617-24. doi: 10.1111/j.1743-6109.2011.02353.x. Epub 2011 Jun 27. PMID 21707928

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil: Tadalafil 5 milligrams (mg) administered orally once a day for 12 weeks. Dosing started at 5 mg tadalafil daily and could be down-titrated to 2.5 mg tadalafil daily based on individual tolerability. (Doses could subsequently be increased back to 5 mg based on response.)
- Placebo: Placebo tablets, matching 5 mg and 2.5 mg tadalafil tablets, given once daily by oral administration for 12 weeks.
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 147 | 70
Completed | 130 | 64
Not Completed | 17 | 6
Not completed — Adverse Event | 4 | 1
Not completed — Sponsor Decision | 0 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 147 | 70 | 217
Age Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.90) | 51.9 (10.35) | 52.1 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 147 | 70 | 217
Race/Ethnicity, Customized [Number; unit: participants]
  White | 144 | 69 | 213
  Asian | 2 | 0 | 2
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Germany | 39 | 19 | 58
  Greece | 19 | 9 | 28
  Italy | 27 | 13 | 40
  Poland | 31 | 14 | 45
  Spain | 31 | 15 | 46
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m²)] | 27.92 (4.685) | 27.74 (3.423) | 27.86 (4.313)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the International Index of Erectile Function - Erectile Function Domain (IIEF-EF) at Week 12
Description: Self-reported erectile function over the past 4 weeks. Scores range from 0 (low or no erectile function) to 5 (high erectile function) on 6 questions (1-5, 15 of the IIEF). Total Erectile Function Domain scores range from 0 to 30.
Time Frame: Baseline, Week 12
Population: The efficacy analysis of the three primary efficacy variables (IIEF-EF, SEP Question 2, and SEP Question 3) was performed on all randomized subjects who had at least one baseline and one post-baseline observation on all three variables.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 67
units on a scale
  Baseline | 15.5 (6.00) | 16.0 (6.27)
  Week 12 Change | 7.3 (6.01) | 3.3 (5.98)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Model included terms for baseline value of efficacy variable, treatment group, country, and the baseline-by-treatment-group interaction. In any model,if the interaction was not significant (if p≥0.10), then the interaction term was removed and the main effects model was used to calculate the between-treatment-group p-value. All tests were based on type 3 sums of squares; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for Week 12 Change. The null hypothesis concerning tadalafil versus placebo was to be rejected if, and only if, the three primary hypotheses (H01, H02, and H03) were all rejected therefore no adjustments for multiple comparisons were made; Change = Endpoint - Baseline; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [2.2 to 5.5], Standard Error of Mean 0.85

2. Primary Outcome: Change From Baseline in Question 2 of the Patient Sexual Encounter Profile (SEP) Diary at Week 12 in Percentage of Yes Responses
Description: Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 2. "Were you able to insert your penis into your partner's vagina?" Data are presented as the mean percentage of yes responses per participant.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 67
percentage of yes responses
  Baseline | 60.1 (38.77) | 59.9 (38.83)
  Week 12 Change | 23.2 (31.92) | 11.6 (25.48)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Change = Endpoint - Baseline; Mean Difference (Final Values) = 11.7, 95% CI 2-sided [5.1 to 18.3], Standard Error of Mean 3.35

3. Primary Outcome: Sexual Encounter Profile (SEP) Diary, Question 3 Change From Baseline to Week 12 in Percentage of Yes Responses
Description: Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 3. "Did your erection last long enough for you to have successful intercourse?" Data are presented as the mean percentage of yes responses per participant.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 67
percentage of yes responses
  Baseline | 28.2 (31.86) | 32.2 (35.93)
  Week 12 Change | 39.4 (34.71) | 19.3 (36.18)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Change = Endpoint - Baseline; Mean Difference (Final Values) = 18.0, 95% CI 2-sided [8.9 to 27.0], Standard Error of Mean 4.60

4. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Nocturnal Penile Tumescence (NPT) Pattern: Number of Erectile Events Per Night
Description: NPT was measured using electrobioimpedance volumetric assessment (NEVA). The NEVA device measures a man's erections during the night. The man wears the device for three nights prior to visit 2 (baseline), visit 5 (end of randomised treatment) and visit 6 (end of follow-up). Data are entered for the 2 nights prior to the visit. During the night the man may have multiple erections. The number of erections is recorded.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: Number of events per night
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
Number of events per night
  Baseline (n=122, n=63) | 2.75 (2.270) | 2.44 (2.002)
  Week 12 Change (n=96, n=49) | -0.11 (2.592) | -0.09 (2.214)

5. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Nocturnal Penile Tumescence (NPT) Pattern: Duration of Erectile Events Per Night
Description: NPT was measured using electrobioimpedance volumetric assessment (NEVA). The NEVA device measures a man's erections during the night. The duration of erections are measured and recorded. Data presented are the duration of erectile events at baseline and the change from baseline to Week 12.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
minutes
  Baseline (n=104, n=56) | 28.487 (14.4791) | 26.372 (11.8969)
  Week 12 Change (n=65, n=33) | -1.553 (16.0073) | -0.398 (12.4585)

6. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Nocturnal Penile Tumescence (NPT) Pattern: Percentage Volumetric Change
Description: NPT was measured using electrobioimpedance volumetric assessment (NEVA). The NEVA device measures a man's erections during the night. The percent of volume change of the penis during erections is measured and recorded for each erection. Data presented are mean percentage of volumetric change from baseline to Week 12.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: percent of volumetric change
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 65 | 33
percent of volumetric change | -5.96 (74.647) | -50.30 (150.321)

7. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Frequency of Spontaneous Morning Erections Captured by Patient Diary
Description: The morning erection diary allows the participant to record whether he experienced an erection on waking. The participant is to complete the morning erection diary every morning during the run-in, treatment and follow-up periods. The percentage of mornings the participant reported an erection is analysed.
Time Frame: Baseline, 12 weeks
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
percent
  Baseline (n=145, n=67) | 31.0 (27.21) | 28.9 (25.74)
  Week 12 Change (n=145, n=66) | 27.5 (25.29) | 11.9 (22.00)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; The change from baseline to endpoint in morning erection percentages was analyzed with an ANCOVA model including terms for baseline value, treatment group, country, age and the baseline-by-treatment-group interaction. In any model, if the interaction was not significant (at p≥0.10), then the interaction term was removed from the model and the main effects model was used to calculate the between-treatment-group p-value. All tests were based on type 3 sums of squares; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12 change. For secondary endpoints, all tests of hypotheses (null hypothesis versus the alternative hypothesis) were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated; Change = Endpoint - Baseline; Mean Difference (Final Values) = 16.2, 95% CI 2-sided [9.5 to 22.8], Standard Error of Mean 3.37

8. Secondary Outcome: The Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire at 12 Week Endpoint
Description: The subject questionnaire consists of 11 questions. Each question is rated on a scale of 0 (extremely low treatment satisfaction) to 4 (extremely high treatment satisfaction). The EDITS summary score will be obtained by adding each individual result for all questions, dividing by the number of questions answered (mean satisfaction score), and multiplying by 25, thus obtaining a score that ranges from 0 (extremely low treatment satisfaction) to 100 (extremely high satisfaction).
Time Frame: Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
units on a scale | 72.8 (20.66) | 52.7 (22.62)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; The models included terms for baseline value of the efficacy variable,treatment group,country, and the baseline-by-treatment-group interaction.In any model, if the interaction was not significant (at p≥0.10), then the interaction term was removed from the model and the main effects model was used to calculate the between-treatment-group p-value. All tests were based on type 3 sums of squares; Test type: Superiority or Other; p > 0.001, ANOVA — p-value is for Week 12 Change. For secondary endpoints, all tests of hypotheses were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated; Mean Difference (Final Values) = 20.0, 95% CI 2-sided [13.9 to 26.1], Standard Error of Mean 3.11

9. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Total and Subdomain Scores of the Self-Esteem and Relationship (SEAR) Questionnaire
Description: SEAR measures improvement in self-esteem and relationship satisfaction. Questionnaire consists of two domains, Sexual Relationship (items 1-8) and Confidence (items 9-14). All questions except negatively worded questions 8 and 11 are scored from 1=almost never/never to 5=almost always/always. Questions 8 and 11 were reverse scored, thus a higher score signifies a more favorable response for all 14 items. Overall score is transformed into a 0 (least favorable) to 100 (most favorable) scale.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
units on a scale
  Total (Baseline) | 47.3 (21.95) | 47.9 (21.58)
  Total (Change) | 20.4 (23.85) | 8.3 (21.14)
  Sexual Relationship Domain (Baseline) | 43.0 (22.54) | 43.9 (21.68)
  Sexual Relationship Domain (Change) | 23.4 (25.88) | 9.7 (22.35)
  Confidence Domain (Baseline) | 53.1 (25.58) | 53.1 (24.85)
  Confidence Domain (Change) | 16.5 (25.58) | 6.5 (24.57)
  Self-Esteem Domain (Baseline) | 50.5 (28.15) | 48.5 (30.06)
  Self-Esteem Domain (Change) | 19.2 (27.85) | 9.3 (30.05)
  Overall Relationship Domain (Baseline) | 58.2 (31.47) | 62.3 (29.01)
  Overall Relationship Domain (Change) | 11.0 (32.51) | 0.9 (30.17)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; The model included terms for baseline value of the efficacy variable, treatment group, country, and the baseline-by-treatment-group interaction. In any model, if the interaction was not significant (at p≥0.10), then the interaction term was removed from the model and the main effects model was used to calculate the between-treatment-group p-value. All tests were based on type 3 sums of squares; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for Total (Change). For secondary endpoints, all tests of hypotheses (null hypothesis versus the alternative hypothesis) were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated; Change = Endpoint - Baseline; Mean Difference (Final Values) = 11.7, 95% CI 2-sided [5.5 to 18.0], Standard Error of Mean 3.17
Statistical Analysis 2: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for Sexual Relationship Domain(Change).For secondary endpoints, all tests of hypotheses (null hypothesis versus the alternative hypothesis) were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated; Change = Endpoint - Baseline; Mean Difference (Final Values) = 13.2, 95% CI 2-sided [6.6 to 19.8], Standard Error of Mean 3.36
Statistical Analysis 3: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0034, ANCOVA — p-value is for Confidence Domain (Change).For secondary endpoints, all tests of hypotheses (null hypothesis versus the alternative hypothesis) were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated; Change = Endpoint - Baseline; Mean Difference (Final Values) = 9.9, 95% CI 2-sided [3.3 to 16.5], Standard Error of Mean 3.34
Statistical Analysis 4: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0020, ANCOVA — p-value is for Self-Esteem Domain (Change).For secondary endpoints, all tests of hypotheses (null hypothesis versus the alternative hypothesis) were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated; Change = Endpoint - Baseline; Mean Difference (Final Values) = 11.0, 95% CI 2-sided [4.1 to 17.9], Standard Error of Mean 3.52
Statistical Analysis 5: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0653, ANCOVA — p-value is for Overall Relationship Domain(Change).For secondary endpoints, all tests of hypotheses (null hypothesis versus the alternative hypothesis) were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated; Change = Endpoint - Baseline; Mean Difference (Final Values) = 7.5, 95% CI 2-sided [-0.5 to 15.6], Standard Error of Mean 4.07

10. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Index of Erectile Function (IIEF), Orgasmic Functions (OF)
Description: Self-reported overall satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction) to 5 (high satisfaction), thus the 2 questions of the IIEF-OF domain range from 0 to 10.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
units on a scale
  Baseline | 6.5 (2.99) | 7.2 (2.81)
  Week 12 Change | 2.0 (2.78) | 0.5 (2.02)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for Week 12 Change.For secondary endpoints, all tests of hypotheses were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated; Change = Endpoint - Baseline; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.7 to 1.9], Standard Error of Mean 0.29

11. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Index of Erectile Function (IIEF), Sexual Desire (SD)
Description: Self-reported overall satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction to 5 (high satisfaction), thus the 2 questions of the IIEF-SD domain range from 0 to 10.
Time Frame: Baseline, 12 weeks
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
units on a scale
  Baseline | 6.7 (1.81) | 6.6 (1.87)
  Week 12 Change | 0.5 (1.93) | -0.1 (1.78)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0089, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Change = Endpoint - Baseline; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [0.2 to 1.1], Standard Error of Mean 0.25

12. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Index of Erectile Function (IIEF), Intercourse Satisfaction (IS)
Description: Self-reported intercourse satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction) to 5 (high satisfaction), thus the 3 questions of the IIEF-IS domain range from 0 to 15.
Time Frame: Baseline, Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
units on a scale
  Baseline | 8.2 (2.65) | 7.6 (2.43)
  Week 12 Change | 2.1 (2.67) | 1.5 (2.56)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0461, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Change = Endpoint - Baseline; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.0 to 1.5], Standard Error of Mean 0.37

13. Secondary Outcome: Change From Baseline to 12 Week Endpoint in International Index of Erectile Function (IIEF), Overall Satisfaction (OS)
Description: Self-reported overall satisfaction over the past 4 weeks. Scores range from 0 (low/no satisfaction to 5 (high satisfaction), thus the 2 questions of the IIEF-OS domain range from 0 to 10.
Time Frame: Baseline, 12 weeks
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
units on a scale
  Baseline | 5.2 (2.15) | 5.1 (2.11)
  Week 12 Change | 2.0 (2.37) | 0.8 (2.19)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Change = Endpoint - Baseline; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.7 to 1.9], Standard Error of Mean 0.30

14. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Sexual Encounter Profile (SEP) Question 1 Percentage of "Yes" Responses
Description: Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 1. "Were you able to achieve at least some erection (some enlargement of the penis)? " Data are presented as the mean percentage of yes responses per participant.
Time Frame: Baseline, 12 weeks
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
percentage of yes responses
  Baseline | 80.8 (28.52) | 74.2 (34.26)
  Week 12 Change | 12.5 (24.03) | 9.5 (24.67)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; The model included terms for baseline value of the efficacy variable, treatment group, country, and the baseline-by-treatment-group interaction. In any model, if the interaction was not significant (that is, if p≥0.10), then the interaction term was removed from the model and the main effects model was used to calculate the between-treatment-group p-value. All tests were based on the type 3 sums of squares; Test type: Superiority or Other; p = 0.0047, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Baseline = Visit 2; Endpoint = the last non-missing post-baseline value until Visit 5; Change = Endpoint - Baseline; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [2.0 to 10.7], Standard Error of Mean 2.22

15. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Sexual Encounter Profile (SEP) Question 4 Percentage of "Yes" Responses
Description: Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 4. "Were you satisfied with the hardness of your erection?" Data are presented as the mean percentage of yes responses per participant.
Time Frame: Baseline, 12 weeks
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
percentage of yes responses
  Baseline | 11.7 (21.16) | 14.6 (23.30)
  Week 12 Change | 44.1 (35.75) | 18.3 (32.14)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Baseline = Visit 2; Endpoint = the last non-missing post-baseline value until Visit 5; Change = Endpoint - Baseline; Mean Difference (Final Values) = 24.5, 95% CI 2-sided [14.6 to 34.3], Standard Error of Mean 4.99

16. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Sexual Encounter Profile (SEP) Question 5 Percentage of "Yes" Responses
Description: Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Question 5. "Were you satisfied overall with this sexual experience?" Data are presented as the mean percentage of yes responses per participant.
Time Frame: Baseline, 12 weeks
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
percentage of yes responses
  Baseline | 10.3 (20.36) | 12.9 (22.11)
  Week 12 Change | 43.2 (35.52) | 18.5 (30.98)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Baseline = Visit 2; Endpoint = the last non-missing post-baseline value until Visit 5; Change = Endpoint - Baseline; Mean Difference (Final Values) = 23.5, 95% CI 2-sided [13.7 to 33.2], Standard Error of Mean 4.96

17. Secondary Outcome: Global Assessment Question (GAQ) Question 1 at 12 Week Endpoint
Description: GAQ Question 1: Choose the one number which best describes how you perceive your ability to achieve and maintain your erections now, compared to how it was before you began taking medication in this study. Responses range from 1=very much better to 7=very much worse.
Time Frame: Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Number; unit: participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
participants
  Very Much Better | 49 (33.6) | 7 (10.1)
  Much Better | 41 (28.1) | 8 (11.6)
  Little Better | 29 (19.9) | 19 (27.5)
  No Change | 14 (9.6) | 24 (34.8)
  A Little Worse | 5 (3.4) | 5 (7.2)
  Much Worse | 4 (1.4) | 3 (4.3)
  Very Much Worse | 2 (1.4) | 1 (1.4)
  Missing | 4 (2.7) | 2 (2.9)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Wilcoxon's rank sum test was used to compare responses to GAQs between treatment groups; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — p-value is for Global Assessment Questions GAQ1. For secondary endpoints, all tests of hypotheses were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated

18. Secondary Outcome: Global Assessment Question (GAQ) Question 2 at 12 Week Endpoint
Description: GAQ Question 2: Choose the one number which best describes how you perceive your sexual life is now, compared to how it was before you began taking medication in this study. Responses range from 1=very much better to 7=very much worse.
Time Frame: Week 12
Population: The ITT analysis set included all randomized subjects who had a baseline and post-baseline observation.
Measure: Number; unit: participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 146 | 69
participants
  Very Much Better | 40 (27.4) | 5 (7.2)
  Much Better | 49 (33.6) | 11 (15.9)
  Little Better | 28 (19.2) | 17 (24.6)
  No Change | 17 (11.6) | 27 (39.1)
  A Little Worse | 3 (2.1) | 4 (5.8)
  Much Worse | 4 | 3
  Very Much Worse | 1 (0.7) | 0 (0)
  Missing | 4 (2.7) | 2 (2.9)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Wilcoxon's rank sum test was used to compare responses to GAQs between treatment groups; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — p-value is for Global Assessment Question GAQ2.For secondary endpoints, all tests of hypotheses were performed as two-sided tests at the 0.05 significance level (α=0.05) unless otherwise stated

ADVERSE EVENTS:
Groups:
- Tadalafil: Tadalafil 5 milligrams administered orally once a day over 12 weeks. Dosing started at 5 mg tadalafil daily (or matching placebo) and could be down-titrated to 2.5 mg tadalafil daily (or matching placebo) based on individual tolerability. (Doses could subsequently be increased back to 5 mg based on response.)
- Placebo: Placebo tablets, matching 5 mg and 2.5 mg tadalafil tablets, given once daily by oral administration.
Arm/Group | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 2/147 | 1/70
Other Adverse Events (participants affected / at risk) | 27/147 | 7/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=147) | Placebo (N=70)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=147) | Placebo (N=70)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Chest pain (General disorders) | 1 (3) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Maxillary antrum operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days